CLINICAL TRIAL: NCT05045300
Title: Paraneural Sheath and Fascial Compartments Surrounding the Brachial Plexus at the Supraclavicular Fossa: A Retrospective Review of High Definition Ultrasound Images Acquired During Selective Trunk Brachial Plexus Blockade
Brief Title: Paraneural Sheath & Fascial Compartments Surround Brachial Plexus at Supraclavicular Fossa During Selective Trunk Block
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof Manoj K Karmakar, Professor, Chinese University of Hong Kong
Other Study IDs: CRE.2021.474
Record Dates: First submitted 2021-08-31; First posted 2021-09-16 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Musculoskeletal Diseases or Conditions
Keywords: Selective Trunk block
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Ultrasound guided Selective trunk block — High definition ultrasound images that were acquired during USG SeTB are routinely stored in the hard disk of ultrasound machine in DICOM (Digital Imaging and Communications in Medicine) format will be used for this review. The images of principal investigator's previous research studies with Clinical trial registration: NCT04752410 and NCT04773405 will also be retrieved. The ultrasound imaging was performed before (scout scan), during and immediately after the USG SeTB. As is the principal investigator's standard practice, all ultrasound scan was performed in a sequential manner (SUIT: Sequential Ultrasound Imaging Technique) with the orientation marker of the transducer directed laterally so as to obtain a transverse oblique view of the brachial plexus block at the supraclavicular fossa. Approximate 50 cases who had undergone USG SeTB for surgical anesthesia during upper extremity surgery since January 1 2020 to June 30, 2021 will be evaluated by two anesthesiologists.
  Other Names: Ultrasound imaging

SUMMARY:
The aim of this retrospective study is to define the paraneural (fascial) sheath and fascial compartments that surround the brachial plexus at the supraclavicular fossa by reviewing previous ultrasound images from cases that have undergone ultrasound guided selective trunk brachial plexus block.

DETAILED DESCRIPTION:
The optimal anatomical plane (relative to the nerve) or the "goal" for local anesthetic (LA) injection during an ultrasound guided (USG) brachial plexus blockade (BPB) at the supraclavicular fossa is currently not known. USG BPB is often described as a "subfascial", "extra fascial", "intracluster", "interfascial", sub-perineural", "intraneural", "corner pocket" or "periplexus" injection. Although this suggests that the local anesthetic is injected into different tissue planes or fascial compartments, even if such planes do exist, as seen in other regions such as popliteal sciatic nerve are not clearly defined at the supraclavicular fossa. However, recently with the use of high definition ultrasound imaging for USG Selective trunk block (SeTB) and principal investigator has often observed distinct paraneural (fascial) sheath and fascial compartments surrounding the brachial plexus at the supraclavicular fossa. These connective tissue layers are also better delineated after the local anesthetic injection. The principal investigator believes these may be the connective tissue layers that previous researchers have referred to in different reports. Currently there are no published data demonstrating the paraneural sheath and fascial compartment surrounding the brachial plexus in-vivo. Principal investigator believes that this fascial layer and compartment influence the spread of LA during USG BPB around the individual elements of the brachial plexus at the supraclavicular fossa and therefore, these anatomical structures have to be delineated so as to improve the safety, success and quality of USG BPB. This study will involve reviewing archived high definition ultrasound images in audio video interleave format from all adult patients who had undergone USG SeTB for surgical anesthesia during upper extremity surgery from January 1, 2020 to June 30, 2021 to define the paraneural sheath and fascial compartments that surround the brachial plexus at the supraclavicular fossa.

ELIGIBILITY:
Inclusion Criteria:

* Archived high definition ultrasound images (datasets) in audio video interleave (AVI) format from all adult patients who had undergone ultrasound guided selective trunk block for surgical anesthesia during upper extremity surgery since the year 2020 (from 01/01/2020 to 30/06/2021).

Exclusion Criteria:

* patients > 75 years old
* American Society of Anesthesiologists (ASA) physical status > Ⅲ
* previous history of surgery at ipsilateral neck.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dataset of previous research titled "Selective Trunk Block: A Prospective Non-Randomized Study of Intervention" (approved by the Joint CUHK-NTEC CREC; CREC Ref no: 2020.687-T; Clinical trial registration: NCT04752410) and " Minimum Effective Local Anaesthetic Volume of a 1:1 Mixture of 2% Lidocaine with 5 µg/ml of Epinephrine and 0.5% Levobupivacaine Required for Ultrasound Guided Selective Trunk Block: A Dose Finding Study" (approved by the Joint CUHK-NTEC CREC; CREC Ref no:2020.680-T; Clinical trial registration: NCT04773405) will also be retrieved.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Visualization of anatomical nerve structures | through study completion, an average of 1 month
  Two anesthesiologists with extensive experience in regional anesthesia and familiar with the fascial anatomy of the brachial plexus at the supraclavicular fossa will independently review the archived ultrasound images and compare the presence of anatomical nerve structures before and after local anesthetic injection. The structure viewed will be scored as 0=no, 1= yes. If a structure is visualized then a previously reported four-point numerical scale, (0=not visible, 1= hardly visible, 2=well visible, 3= very well visible_ will be used to assess the quality of ultrasound visibility. The total ultrasound visibility score (UVS) of the anatomical structures in the transverse scan will be calculated for every subject (maximum score possible = 30) and the mean total UVS will be determined by averaging the scores of the two observers. Inter-rater agreement of the aforementioned anatomical structures between the anesthesiologist will be calculated using kappa statistics.

SECONDARY OUTCOMES:
Visualization of the presence of anatomical variations | through study completion, an average of 1 month
  Two anesthesiologists with extensive experience in regional anesthesia and familiar with the fascial anatomy of the brachial plexus at the supraclavicular fossa will independently review the archived ultrasound images and compare the presence of anatomical variations before and after local anesthetic agent injection. It will be scored as 0=not presence, 1=presence.
Presence of artery within the nerve cluster | through study completion, an average of 1 month
  Two anesthesiologists with extensive experience in regional anesthesia and familiar with the fascial anatomy of the brachial plexus at the supraclavicular fossa will independently review the archived ultrasound images and evaluate the presence or absence of blood vessels inside the nerve cluster at the supraclavicular fossa. A score of 0=not presence and 1=presence.

CONTACTS AND LOCATIONS:
Overall Officials: Manoj K Karmakar, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Anaesthesia & Intensive Care, Prince of Wales Hospital, Shatin, New Territories, Hong Kong